CLINICAL TRIAL: NCT00411450
Title: Multi Center, Open Label, Single Arm Trial Evaluating Panitumumab in Combination With FOLFIRI Therapy Following First Line FOLFOX and Bevacizumab Treatment of Metastatic Colorectal Cancer
Brief Title: Panitumumab Regimen Evaluation in Colorectal Cancer to Estimate Primary Response to Treatment
Acronym: PRECEPT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20060277
Record Dates: First submitted 2006-12-12; First posted 2006-12-14 (Estimated); Results first posted 2016-02-15 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-01

CONDITIONS: Colon Cancer; Colorectal Cancer; Rectal Cancer; Cancer; Metastatic Cancer; Metastatic Colorectal Cancer; Oncology
Keywords: k-ras; biomarker; colorectal; colon; rectal; FOLFOX; FOLFIRI
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Rectal Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — Panitumumab; IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Panitumumab plus FOLFIRI (Experimental): Participants received 6 mg/kg panitumumab intravenously (IV) once every 14 days in combination with FOLFIRI chemotherapy regimen consisting of irinotecan, infusional 5-fluorouracil, and leucovorin, until disease progression, intolerability, death, or study withdrawal.
  Interventions: Biological: Panitumumab; Drug: FOLFIRI

INTERVENTIONS:
Biological: Panitumumab — Administered by intravenous infusion
  Other Names: Vectibix
Drug: FOLFIRI — Chemotherapy consisting of irinotecan with infusional 5-fluorouracil and leucovorin. Recommended dosage regimen and administration of FOLFIRI was based on local standard of care, the package insert for each product, and institutional guidelines.

SUMMARY:
The primary objective is to estimate the effect of the human homolog of the Kirsten rat sarcoma-2 virus oncogene (KRAS) mutation status (wild type versus mutant) from tumor tissue on efficacy endpoints in patients with metastatic colorectal cancer (mCRC) receiving second-line chemotherapy with panitumumab after failing first-line treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic adenocarcinoma of the colon or rectum
* Available paraffin-embedded tumor tissue
* Failure of first line treatment containing fluoropyrimidine and oxaliplatin based chemotherapy with bevacizumab for mCRC
* Measurable disease
* Adequate hematologic, renal, hepatic and metabolic function

Exclusion Criteria:

* Radiotherapy ≤ 2 weeks prior to Day 1 of Cycle 1
* Unresolved toxicity(ies) from prior anti cancer therapy that, in the opinion of the investigator, precludes the subject from study enrollment
* Prior irinotecan therapy, anti epidermal growth factor receptor (EGFr) therapy, or vaccine for the treatment of mCRC
* CYP3A4 enzyme inducers, inhibitors, and substrates (eg, phenytoin, phenobarbital, carbamazepine, ketoconazole, rifampin, rifabutin, and St. John's Wort) ≤ 2 weeks prior to Day 1 of Cycle 1
* Infection requiring systemic anti infectives completed ≤ 2 weeks prior to Day 1 of Cycle 1
* Clinically significant cardiovascular disease
* History of interstitial lung disease (eg, pneumonitis or pulmonary fibrosis)
* Pulmonary embolism, deep vein thrombosis, or other significant thromboembolic event ≤ 8 weeks prior to Day 1 of Cycle 1
* Any significant bleeding ≤ 6 weeks prior to Day 1 of Cycle 1, per the investigator's judgement
* Gastroduodenal ulcer(s) determined by endoscopy to be active or uncontrolled gastrointestinal ulcer ≤ 4 weeks prior to Day1 of Cycle 1
* Any co-morbid disease or condition that could increase the risk of toxicity (eg, dihydropyrimidine deficiency, significant ascites, or pleural effusion)
* Major surgery (requiring general anesthesia), open biopsy, or significant traumatic injury ≤ 4 weeks prior to Day1 of Cycle 1. Subjects must have recovered from surgery and have no significant complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2006-11; Primary Completion 2009-01 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Cohn AL, Shumaker GC, Khandelwal P, Smith DA, Neubauer MA, Mehta N, Richards D, Watkins DL, Zhang K, Yassine MR. An open-label, single-arm, phase 2 trial of panitumumab plus FOLFIRI as second-line therapy in patients with metastatic colorectal cancer. Clin Colorectal Cancer. 2011 Sep;10(3):171-7. doi: 10.1016/j.clcc.2011.03.022. Epub 2011 Apr 28. PMID 21855038
- [Derived] Weeraratne D, Chen A, Pennucci JJ, Wu CY, Zhang K, Wright J, Perez-Ruixo JJ, Yang BB, Kaliyaperumal A, Gupta S, Swanson SJ, Chirmule N, Starcevic M. Immunogenicity of panitumumab in combination chemotherapy clinical trials. BMC Clin Pharmacol. 2011 Nov 9;11:17. doi: 10.1186/1472-6904-11-17. PMID 22070868
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 56 sites in the United States. The first patient enrolled on 30 November 2006 and the last patient enrolled on 07 January 2008.
Pre-assignment Details: Participants recived second-line therapy until disease progression, intolerability, death, or study withdrawal. Participants completed a safety visit 4 weeks after the last dose. Participants were followed for survival every 12 weeks from the safety visit until the end of the study; the data cut-off date for results is 2 January 2009.
Period: Overall Study
Arm/Group | Panitumumab Plus FOLFIRI
Started | 116
Received Treatment | 115
Completed | 113 (Ended second-line treatment)
Not Completed | 3
Not completed — Ongoing at time of data cut-off. | 3

BASELINE CHARACTERISTICS:
Arm/Group | Panitumumab Plus FOLFIRI
Number analyzed (Participants) | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 75
Race/Ethnicity, Customized [Number; unit: participants]
  White or Caucasian | 94
  Black or African American | 13
  Hispanic or Latino | 8
  Asian | 1
Kirsten Rat Sarcoma Gene (KRAS) Mutation Status [Number; unit: participants] — Unevaluable includes missing, lack of tissue sample, invalid or failed test results.
  participants
    Wild-type | 65
    Mutant | 45
    Unevaluable | 6

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate at Weeks 17 and 25
Description: Objective response rate is defined as the percentage of participants with a best response of complete response or partial response. Disease assessments were based on investigator review of scans using modified Response Evaluation Criteria in Solid Tumors (RECIST) criteria. A complete or partial response was confirmed no less than 4 weeks after the criteria for response were first met. Participants with no radiographic tumor assessment(s) at Week 17 or 25 were considered non-responders. Complete Response (CR): disappearance of all target and non-target lesions and no new lesions. Partial Response (PR): At least a 30% decrease in the size of target lesions with no progression of non-target lesions (defined as a ≥ 25% increase in lesion size) and no new lesions, or, the disappearance of all target lesions but persistence of 1 or more non-target lesions not qualifying for either CR or progressive disease (PD) and no new lesions.
Time Frame: Week 17 and Week 25
Population: Tumor Response Analysis Set (all participants who provided informed consent prior to the initiation of any study specific procedures, received at least 1 dose of panitumumab, who had valid KRAS mutation status data available and with at least 1 uni-dimensionally measurable lesion per the local investigator)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Wild-type KRAS: Participants with wild-type KRAS received 6 mg/kg panitumumab intravenously (IV) once every 14 days in combination with FOLFIRI chemotherapy regimen consisting of irinotecan, infusional 5-fluorouracil, and leucovorin.
- Mutant KRAS: Participants with mutant KRAS received 6 mg/kg panitumumab intravenously (IV) once every 14 days in combination with FOLFIRI chemotherapy regimen consisting of irinotecan, infusional 5-fluorouracil, and leucovorin.
Arm/Group | Wild-type KRAS | Mutant KRAS
Number analyzed (Participants) | 64 | 43
percentage of participants
  Week 17 | 20 [10 to 30] | 14 [4 to 24]
  Week 25 | 22 [12 to 32] | 14 [4 to 24]
Statistical Analysis 1: Comparison: Wild-type KRAS vs Mutant KRAS; Difference at Week 17; Test type: Superiority or Other; Difference = 6, 95% CI 2-sided [-11 to 21] — Difference = Wild type - Mutant
Statistical Analysis 2: Comparison: Wild-type KRAS vs Mutant KRAS; Difference at Week 25; Test type: Superiority or Other; Difference = 8, 95% CI 2-sided [-9 to 23]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: The severity of adverse events (AEs) was graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0, except for panitumumab related skin toxicities, where Grade 1 = Mild AE; Grade 2 = Moderate AE; Grade 3 = Severe AE; Grade 4 = Life-threatening or disabling AE; Grade 5 = Death related to AE. The relationship of each adverse event to the panitumumab and/or FOLFIRI regimen was assessed by the investigator. A serious adverse event was defined as an adverse event that • is fatal • is life threatening • requires in-patient hospitalization or prolongation of existing hospitalization • results in persistent or significant disability/incapacity • is a congenital anomaly/birth defect • other significant medical hazard.
Time Frame: From the first dose date to 30 days after the last dose date. The median time frame is 4.5 months.
Population: Safety analysis set (all participants who provided informed consent prior to the initiation of any study specific procedure and who received at least 1 dose of panitumumab)
Measure: Number; unit: participants
Arm/Group | Panitumumab Plus FOLFIRI
Number analyzed (Participants) | 115
participants
  Any adverse event | 115
  Grade 3 or higher adverse event | 94
  Panitumumab-related adverse events | 107
  Chemotherapy-related adverse events | 112
  ≥ grade 3 panitumumab-related adverse events | 56
  ≥ grade 3 chemotherapy-related adverse events | 65
  Serious adverse events | 46
  Serious panitumumab-related adverse events | 15
  Serious chemotherapy-related adverse events | 24
  Life-threatening adverse events | 18
  Ended second-line treatment due to adverse events | 18
  Ended panitumumab due to adverse events | 20
  Ended FOLFIRI due to adverse events | 28
  Death due to adverse events | 8
  Panitumumab infusion reactions | 2
  Deaths during study | 71

3. Primary Outcome: Best Response During Second-Line Treatment
Description: Objective response rate is defined as the percentage of participants with a best response of complete response or partial response based on investigator review of scans using modified RECIST criteria. A complete or partial response was confirmed no less than 4 weeks after the criteria for response were first met. Participants with no post-baseline radiographic tumor assessment(s) were considered non-responders.
  CR: disappearance of all target and non-target lesions and no new lesions. PR: At least a 30% decrease in the size of target lesions with no progression of non-target lesions (defined as a ≥ 25% increase in lesion size) and no new lesions, or, the disappearance of all target lesions but persistence of 1 or more non-target lesions not qualifying for either CR or PD and no new lesions.
Time Frame: Tumor response was assessed at Weeks 9, 17, 25, and 33, and once every 12 weeks thereafter until the end of second-line treatment; maximum time on treatment was 77 weeks.
Population: Tumor Response Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Wild-type KRAS | Mutant KRAS
Number analyzed (Participants) | 64 | 43
percentage of participants | 23 [13 to 34] | 16 [5 to 27]
Statistical Analysis 1: Comparison: Wild-type KRAS vs Mutant KRAS; Test type: Superiority or Other; Difference = 7, 95% CI 2-sided [-11 to 23] — Difference = Wild type - Mutant

4. Primary Outcome: Progression-free Survival Rate at Weeks 17 and 25
Description: The progression-free survival rate is defined as the Kaplan-Meier (KM) estimator of progression-free survival at Week 17 and Week 25 reported as the probability of being event (disease progression or death)-free. Tumor assessments were evaluated by the investigator according to modified RECIST criteria.
  PD: At least a 20% increase in the size of target lesions since the treatment started or at least a 25% increase in the size of non-target lesions and the lesion(s) measure ≥ 10 mm, or the appearance of any new lesions. Participants who withdraw from the study prior to completion of Week 17 or 25 radiographic tumor assessments were censored at the last evaluable tumor assessment.
Time Frame: Week 17 and Week 25
Population: Primary Analysis Set (all participants who provided informed consent prior to the initiation of any study specific procedures, received at least 1 dose of panitumumab, and who had valid KRAS mutation status data available)
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Wild-type KRAS | Mutant KRAS
Number analyzed (Participants) | 64 | 45
percent probability
  Week 17 | 67 [54 to 77] | 55 [39 to 68]
  Week 25 | 52 [39 to 64] | 41 [27 to 55]
Statistical Analysis 1: Comparison: Wild-type KRAS vs Mutant KRAS; Difference at Week 17; Test type: Superiority or Other; Difference = 12.5, 95% CI 2-sided [-6.3 to 31.4] — Difference = Wild type - Mutant
Statistical Analysis 2: Comparison: Wild-type KRAS vs Mutant KRAS; Difference at Week 25; Test type: Superiority or Other; Difference = 10.9, 95% CI 2-sided [-8.4 to 30.2]

5. Primary Outcome: Progression-free Survival Time
Description: Progression-free survival time was defined as the time from Study Day 1 to the date of disease progression (based on investigator assessment) or the date of death due to any cause. Participants who terminated from the study early (eg, prior to disease progression due to fully withdrawn informed consent) were censored at their last tumor assessment.
Time Frame: From Study Day 1 until the data cut-off date of 2 January 2009; median follow-up time was 39 weeks, with a maximum of 93 weeks.
Population: Primary Analysis Set
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Wild-type KRAS | Mutant KRAS
Number analyzed (Participants) | 64 | 45
weeks | 26 [19 to 33] | 19 [12 to 25]
Statistical Analysis 1: Comparison: Wild-type KRAS vs Mutant KRAS; Test type: Superiority or Other; Hazard Ratio (HR) = 0.8, 95% CI 2-sided [0.5 to 1.1] — Hazard ratio estimated from a Cox Proportional Hazards regression model with only KRAS effect (Wild type vs. Mutant)

6. Primary Outcome: Disease Control Rate at Weeks 17 and 25
Description: The percentage of participants whose best response was either a complete or partial response or stable disease, based on modified RECIST criteria as assessed by the investigator. Stable diease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD of target lesions and no progression of existing non-target lesions and no new lesions, or, the persistence of 1 or more non-target lesions not qualifying for either CR or PD if no target lesions were identified at Baseline.
Time Frame: Week 17 and Week 25
Population: Tumor Response Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Wild-type KRAS | Mutant KRAS
Number analyzed (Participants) | 64 | 43
percentage of participants
  Week 17 | 64 [52 to 76] | 58 [43 to 73]
  Week 25 | 64 [52 to 76] | 58 [43 to 73]
Statistical Analysis 1: Comparison: Wild-type KRAS vs Mutant KRAS; Difference at Week 17; Test type: Superiority or Other; Difference = 6, 95% CI 2-sided [-14 to 25] — Difference = Wild type - Mutant
Statistical Analysis 2: Comparison: Wild-type KRAS vs Mutant KRAS; Difference at Week 25; Test type: Superiority or Other; Difference = 6, 95% CI 2-sided [-14 to 25]

7. Primary Outcome: Duration of Response
Description: Duration of response is defined as the time from the date of first response to the date of first progression of disease during second-line treatment (as evaluated by the investigator) or death (if the death was due to disease progression but not detected earlier) in the subset of participants who responded (CR or PR, as evaluated by the investigator). Duration of response was analyzed using Kaplan-Meier methods; participants who responded but did not progress while on study were censored at the date of last tumor assessment.
Time Frame: as for outcome 3
Population: Responders of Tumor Response Analysis Set
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Wild-type KRAS | Mutant KRAS
Number analyzed (Participants) | 15 | 7
weeks | 29 [21 to 39] | 23 [16 to 74]
Statistical Analysis 1: Comparison: Wild-type KRAS vs Mutant KRAS; Test type: Superiority or Other; Hazard Ratio (HR) = 0.7, 95% CI 2-sided [0.2 to 2.0] — Hazard ratio estimated from a Cox Proportional Hazards regression model with only KRAS effect (Wild type vs. Mutant)

8. Primary Outcome: Overall Survival
Description: Overall survival is defined as as the number of days from Study Day 1 to the date of death due to any cause. Overall survival was analyzed using the Kaplan-Meier method; participants who were lost to follow-up or who had not died at the end of the study (52 weeks after the last participant was enrolled) were censored at the date of last contact.
Time Frame: as for outcome 5
Population: Primary Analysis Set
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Wild-type KRAS | Mutant KRAS
Number analyzed (Participants) | 64 | 45
weeks | 50 [39 to 76] | 31 [23 to 47]
Statistical Analysis 1: Comparison: Wild-type KRAS vs Mutant KRAS; Test type: Superiority or Other; Hazard Ratio (HR) = 0.6, 95% CI 2-sided [0.4 to 0.9] — Hazard ratio estimated from a Cox Proportional Hazards regression model with only KRAS effect (Wild type vs. Mutant)

9. Primary Outcome: Time to Treatment Failure
Description: Time to failure of second-line treatment is defined as the time from study Day 1 to the date of the earliest of the following events: end of second-line therapy due to any reason except for complete response and curative surgery; progressive disease; or death due to any cause. Time to treatment failure was analyzed using Kaplan-Meier methods; participants who did not discontinue second-line treatment or discontinue due to complete response or curative surgery, who were still alive, and who did not have disease progression were censored at the date of the last contact.
Time Frame: as for outcome 3
Population: Primary Analysis Set
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Wild-type KRAS | Mutant KRAS
Number analyzed (Participants) | 64 | 45
weeks | 19 [14 to 25] | 15 [8 to 19]
Statistical Analysis 1: Comparison: Wild-type KRAS vs Mutant KRAS; Test type: Superiority or Other; Hazard Ratio (HR) = 0.7, 95% CI 2-sided [0.5 to 1.1] — Hazard ratio estimated from a Cox Proportional Hazards regression model with only KRAS effect (Wild type vs. Mutant)

10. Primary Outcome: Time to Progression
Description: Time to progression is defined as the time from study Day 1 to the date of observed disease progression. Time to progression was analyzed using Kaplan-Meier methods; participants who did not have disease progression were censored at the date of last evaluable tumor assessment.
Time Frame: as for outcome 5
Population: Primary Analysis Set
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Wild-type KRAS | Mutant KRAS
Number analyzed (Participants) | 64 | 45
weeks | 26 [16 to 34] | 17 [15 to 25]
Statistical Analysis 1: Comparison: Wild-type KRAS vs Mutant KRAS; Test type: Superiority or Other; Hazard Ratio (HR) = 0.8, 95% CI 2-sided [0.5 to 1.2] — Hazard ratio estimated from a Cox Proportional Hazards regression model with only KRAS effect (Wild type vs. Mutant)

11. Primary Outcome: Time to Response
Description: Time to response of second-line treatment is defined as the time from study Day 1 to the date of first documentation of CR or PR, calculated for those participants with an objective tumor response of CR or PR.
Time Frame: as for outcome 3
Population: Responders in the Tumor Response Analysis Set
Measure: Median (Full Range); unit: weeks
Arm/Group | Wild-type KRAS | Mutant KRAS
Number analyzed (Participants) | 15 | 7
weeks | 9.1 [6.9 to 32.3] | 9.3 [7.0 to 35.6]

12. Secondary Outcome: Number of Participants With Grade 4 Laboratory Toxicities
Description: Laboratory toxicities were graded according to CTCAE version 3.
Time Frame: From the first dose date to 30 days after the last dose date. The median time frame is 4.5 months.
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | Panitumumab Plus FOLFIRI
Number analyzed (Participants) | 115
participants
  Anemia | 1
  Neutropenia | 4
  Hypomagnesaemia | 8
  Hypokalemia | 1
  Hypocalcaemia | 3
  Hyperbilirubinaemia | 1

13. Secondary Outcome: Number of Participants Who Developed Antibodies to Panitumumab
Description: The immunogenicity of panitumumab was evaluated using 2 different screening immunoassays for the detection of anti-panitumumab antibodies: an acid dissociation bridging enzyme-linked immunosorbent assay (ELISA; detecting high-affinity antibodies) and a Biacore® biosensor immunoassay (detecting both high and low-affinity antibodies). When either of the 2 screening assays yielded a positive result, that particular sample was subjected to an in vitro bioassay for the detection of neutralizing antibodies.
Time Frame: Prior to first dose and 28 days after the last dose of second-line treatment
Population: Safety Analysis Set with baseline anti-panitumumab antibody testing sample available
Measure: Number; unit: participants
Arm/Group | Panitumumab Plus FOLFIRI
Number analyzed (Participants) | 113
participants
  Binding antibody positive | 1
  Neutralizing antibody positive | 0

ADVERSE EVENTS:
Time Frame: The time frame for adverse event reporting is from the first dose date to 30 days since the last dose date. The median time frame is 4.5 months.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Panitumumab + FOLFIRI: Participants received 6 mg/kg panitumumab intravenously (IV) once every 14 days in combination with FOLFIRI chemotherapy regimen consisting of irinotecan, infusional 5-fluorouracil, and leucovorin, until disease progression, intolerability, death, or study withdrawal.
Arm/Group | Panitumumab + FOLFIRI
Serious Adverse Events (participants affected / at risk) | 46/115
Other Adverse Events (participants affected / at risk) | 114/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab + FOLFIRI (N=115)
Anaemia (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 4
Pancytopenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Atrial fibrillation (Cardiac disorders) | 1
Atrial tachycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Adrenocortical insufficiency acute (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Ileus (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 3
Gait disturbance (General disorders) | 1
Mucosal inflammation (General disorders) | 4
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 6
Hepatic failure (Hepatobiliary disorders) | 1
Abdominal abscess (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Neutropenic sepsis (Infections and infestations) | 1
Perirectal abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 4
Staphylococcal sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 12
Failure to thrive (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Amnesia (Nervous system disorders) | 1
Haemorrhagic stroke (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Sedation (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 3
Anxiety (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 4
Hypotension (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab + FOLFIRI (N=115)
Anaemia (Blood and lymphatic system disorders) | 30
Neutropenia (Blood and lymphatic system disorders) | 33
Thrombocytopenia (Blood and lymphatic system disorders) | 6
Conjunctivitis (Eye disorders) | 6
Lacrimation increased (Eye disorders) | 7
Vision blurred (Eye disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 29
Abdominal pain upper (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 26
Diarrhoea (Gastrointestinal disorders) | 85
Dry mouth (Gastrointestinal disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 64
Stomatitis (Gastrointestinal disorders) | 33
Vomiting (Gastrointestinal disorders) | 34
Asthenia (General disorders) | 12
Catheter thrombosis (General disorders) | 6
Fatigue (General disorders) | 61
Mucosal inflammation (General disorders) | 38
Oedema peripheral (General disorders) | 24
Pain (General disorders) | 10
Pyrexia (General disorders) | 21
Paronychia (Infections and infestations) | 10
Upper respiratory tract infection (Infections and infestations) | 7
Urinary tract infection (Infections and infestations) | 10
International normalised ratio increased (Investigations) | 6
Neutrophil count decreased (Investigations) | 6
Weight decreased (Investigations) | 28
Anorexia (Metabolism and nutrition disorders) | 38
Decreased appetite (Metabolism and nutrition disorders) | 10
Dehydration (Metabolism and nutrition disorders) | 21
Hypokalaemia (Metabolism and nutrition disorders) | 22
Hypomagnesaemia (Metabolism and nutrition disorders) | 23
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 19
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11
Dizziness (Nervous system disorders) | 20
Dysgeusia (Nervous system disorders) | 15
Headache (Nervous system disorders) | 6
Neuropathy peripheral (Nervous system disorders) | 7
Anxiety (Psychiatric disorders) | 13
Depression (Psychiatric disorders) | 8
Insomnia (Psychiatric disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 9
Alopecia (Skin and subcutaneous tissue disorders) | 32
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 44
Dry skin (Skin and subcutaneous tissue disorders) | 28
Erythema (Skin and subcutaneous tissue disorders) | 7
Nail disorder (Skin and subcutaneous tissue disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 24
Rash (Skin and subcutaneous tissue disorders) | 60
Skin fissures (Skin and subcutaneous tissue disorders) | 17
Hypotension (Vascular disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.